CLINICAL TRIAL: NCT03057522
Title: The Effect of a Home Training Program on Preferred Step Rate in Recreational Runners
Brief Title: Step Rate in Recreational Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jonathan T. Finnoff, Professor of Physical Medicine and Rehabilitation, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 16-008532
Record Dates: First submitted 2017-02-14; First posted 2017-02-20 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Gait Disorder, Sensorimotor
Keywords: Run; Cadence; Home exercise
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled study evaluating whether a home exercise program can increase the running cadence of recreational runners.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This group will undergo home exercise program designed to increase their running cadence.
  Interventions: Behavioral: Change in running cadence
- Control Group (No Intervention): This group will not receive any intervention.

INTERVENTIONS:
Behavioral: Change in running cadence — The intervention will involve a home exercise program designed to increase the running cadence in recreational runners.
  Arms: Intervention Group

SUMMARY:
This will be a pilot study to determine if a 6 week home training program can increase preferred step rate (cadence) in recreational runners. Increase in step rate has been correlated with decreased stress at lower limb joints in runners. This has the potential of decreasing overuse injuries in this population.

Research participants will have their preferred cadence evaluated at the beginning of the study. The athletes will be randomly assigned to two groups. One group will continue to train without intervention and the other group will train at a cadence of 10% higher than their preferred step rate.

At the end of 6 weeks the participants will have their preferred cadence reevaluated using the same method as pre-participation cadence was determined.

The investigators hypothesis the preferred running cadence of recreational runners following the intervention will be 5-10% greater than prior to the intervention and the increased cadence will be maintained for 6 months following the intervention.

ELIGIBILITY:
Inclusion criteria:

* healthy male or female runners
* 18 years of age or greater
* run two or more times per week most weeks of the year for at least 4 years
* cadence of 85 strides/min or less as determined at initial evaluation
* no musculoskeletal injuries or illnesses that would limit running in the last 6 months
* currently running at least 15 miles a week

Exclusion criteria:

* baseline running cadence greater than 85 strides/min
* inability to run
* cardiovascular disease
* greater than 2 cardiovascular risk factors
* peripheral vascular disease
* neurological disease
* musculoskeletal injury or disease that causes pain with running

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Running cadence | 6 weeks
  Running cadence (steps per minute) will be evaluated using a running cadence sensor to determine if the intervention subjects increased their running cadence by 10 steps per minute following the intervention.
Running cadence | 6 months
  Running cadence (steps per minute) will be evaluated using a running cadence sensor to determine if the intervention subjects maintained their increased running cadence for 6 months following the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan T Finnoff, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers